CLINICAL TRIAL: NCT00939328
Title: S0902, Phase II Study of Bendamustine Plus Rituximab for the Treatment of Refractory B-Cell Chronic Lymphocytic Leukemia
Brief Title: S0902 Bendamustine and Rituximab in Treating Patients With B-Cell Chronic Lymphocytic Leukemia That Has Not Responded to Previous Treatment
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: question was no longer committee priority
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: S0902; S0902 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Leukemia
Keywords: B-cell chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: rituximab
Drug: bendamustine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as bendamustine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer cell growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cell-killing substances to them. Giving bendamustine together with rituximab may kill more cancer cells.

PURPOSE: This phase II trial is studying the side effects of giving bendamustine together with rituximab and to see how well it works in treating patients with B-cell chronic lymphocytic leukemia that has not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

* To test whether the response rate (CR, CRi, or PR) in patients with purine analog-refractory, B-cell chronic lymphocytic leukemia (CLL) after treatment with the combination of bendamustine hydrochloride and rituximab is sufficiently high to warrant further investigation.
* To evaluate the safety and tolerability of bendamustine hydrochloride and rituximab in patients with B-cell CLL who are refractory to treatment with a purine-nucleoside analog-containing regimen.
* To investigate, in a preliminary manner, the prognostic effects of pre-treatment cytogenetic abnormalities identified by conventional cytogenetics and by FISH analyses on response to treatment in this patient population.

OUTLINE: This is a multicenter study.

Patients receive rituximab IV on day 1 and bendamustine IV over 30 minutes on days 1-2. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. In course 1 only, patients also receive rituximab IV on day 2.

After completion of study treatment, patients are followed up periodically for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically and immunophenotypically confirmed diagnosis of B-cell chronic lymphocytic leukemia (CLL)

  * Progressive or symptomatic disease
  * Purine analog-refractory disease
* Must meet 1 of the following criteria:

  * Intermediate- or high-risk modified-Rai stage
  * Low-risk modified-Rai stage and progressive lymphocytosis, defined as > 50% increase of absolute peripheral lymphocyte count over the lowest count during the past 2 months
* Received 1 or more prior therapies for CLL
* Must be registered on SWOG-9007, "Cytogenetic Studies in Leukemia Patients"

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-3
* ANC > 1,000/mm³
* Platelet count > 50,000/mm³
* Serum creatinine ≤ 2 times upper limit of normal (ULN) OR creatinine clearance ≥ 50 mL/min
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No systemic fungal, bacterial, viral, or other infection that is not controlled (i.e., exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
* No other prior malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for 5 years
* HIV positivity allowed provided the following criteria are met:

  * CD4 cells > 350/mm³
  * No concurrent antiretroviral therapy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 28 days since prior chemotherapy, any other investigational agents, or major surgery
* More than 120 days since prior allogeneic or autologous hematopoietic stem cell transplantation

  * If prior allogeneic bone marrow transplantation, must meet the following criteria:

    * Performed > 120 days ago
    * No acute graft-vs-host disease (GVHD) ≥ grade 2
    * Receiving no immunosuppressive therapy for chronic GVHD
* No concurrent antiretroviral therapy for HIV-positive patients
* No concurrent CYP1A2 inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Response rate (CR, CRi, or PR)
Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Matt E. Kalaycio, MD, Study Chair — The Cleveland Clinic